CLINICAL TRIAL: NCT04491110
Title: Intervention to Improve Sleep Quality in Caregivers of Palliative Care Patients in the Community: Clinical Trial
Brief Title: Intervention to Improve Quality of Sleep of Palliative Patient Carers in the Community: Clinical Trial
Acronym: IMECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Andaluz Health Service (Other Government)
Collaborators: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Principal Investigator, Francisco Javier Navarro Moya, BSc Nursing, Andaluz Health Service
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AP-0225-2019
Record Dates: First submitted 2020-07-13; First posted 2020-07-29 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: Music Therapy; Caregivers; Sleep; Palliative Care
Keywords: Sleep; Caregivers; Music Therapy; Palliative Care; Nurses; Exercise; Physical Exertion
MeSH Terms: conditions — Motor Activity | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: The masking is performed by assigning a mobile phone with headphones and an accelerometer to the carers of the control and intervention group and with the instruction not to mention what they heard to the evaluator; in this sense the participants do not know if they belong to the control or intervention group. However those who listen to music can conclude that it is an intervention group by themselves.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Carer music. (Experimental): Listening to pre-recorded and selected music preferred by the carer, half an hour for 7 days.
  Interventions: Other: Music Therapy
- Sham Comparator: Carer. (Sham Comparator): Basic therapeutic education repetition performed to all carer through earphones, half an hour for 7 days.
  Interventions: Other: simulation with therapeutic education

INTERVENTIONS:
Other: Music Therapy — We are aiming to use music therapy, with pre-recorded favoured music, as a complementary treatment in oncological patients in palliative care, as well as on the carer. It will be done by using mobile telephones.
  Arms: Experimental: Carer music.
Other: simulation with therapeutic education — Basic therapeutic education repetition performed to all caregivers and oncological patients in palliative care, through mobile phones.
  Arms: Sham Comparator: Carer.

SUMMARY:
Introduction Sleeping problems experienced by cancer patients carers are frequent with 72% of carers reporting moderate to severe problems. Another consequence for this carers is the increase of suffering from depression and it is usually associated to carer overload.

Objectives

Main objective:

- To evaluate the effects of listening to music in sleep quality for oncology patients non-professional carers at home, and to evaluate the influence of specific factors that may modify that effect.

Secondary objectives:

* To assess the relationship between the waking state and the consequences during the day according to sleep characteristics. These include:

  1. Psychological results:
  1. Quality of life.
  2. Carer overload.

  2. Physical results:
  1. Sleepiness during the day.
  2. Physical activity, intensity and length evaluation.
* To assess carers satisfaction with the intervention.

Method Randomized clinical trial, single blinding and performed in oncological patients carers in several practices. 2 samples of 40 carers. Intervention group will be taken through a seven session intervention with music; control group will undergo seven sessions of therapeutic education (as a reminder). Results will be evaluated using Pittsburgh Quality of Sleep Index, triaxial accelerometer, EuroQol-5D-5L, Caregiver Strain Index, Epworth Sleepiness Scale and Client Satisfaction Questionnaire.

Statistical analysis Basal values will be compared for both groups. Then the values before and after the intervention will be compared using Student's t distribution for normal continuous variables, and Wilcoxon's T test for paired data in continuous not normal variables. A multiple linear regression will be carried out.

The system developed for the PREDIMEDPLUS study will be used to process accelerometer data results. This semi-automated system manages data capture in a continuous stream in a central server of Malaga University. Processing and analysis of this data is also centralised, with an open source package, GGIR v. 1.5-1248

DETAILED DESCRIPTION:
BACKGROUND AND CURRENT STATUS

Sleep is a complex vital process in which humans spend a third of our lives. Insomnia is related to discontent with quality, length or continuity in that sleep, usually seen as problems to fall sleep, waking up frequently or a sleep that doesn't leave us rested. Progressive shortening on sleep length is a risk factor on developing obesity, diabetes, hypertension, cardiac related conditions and cerebrovascular accident, and can lead to premature death.

Insomnia affects work performance: in severe cases it may lead to a reduction in care or reflexes, increased risk of being involved in accidents, poor morale or social relationships, absence from work and quality of life and immunity reduction.

Regarding sleep decrease in informal carers it is observed that during the condition progress there are several changes in the patients. These changes are related to an increase on sleep alterations in carers, with a mayor prevalence (42 to 95%) in carers of patients with late stage cancer, compared to early stage patients carer (36 to 80%).

Another aspect that may be overlooked frequently is physical activity conducted by carers as a health preventive measure, due to the benefits that physical exercise reports on the health and well-being, including a reduction on risk factors for cardiovascular diseases, cancer, stress and depression reduction, carer overload, mental and cognitive health, and general well-being. Sleep quality improves when physical activity increases in carers.

Insomnia treatment is currently based in pharmaceutical treatment, including sedatives and hypnotic drugs which can provoke dependency and tolerance, reducing their efficacy. These drugs can induce cognitive and behavioural changes, and can lead to severe if not uncommon consequences. Other non-drug related treatments have been developed to deal with insomnia, including music therapy as this induces emotional responses in people. These responses are classified according to good or bad, and also in their intensity, being high or low.

Several theories have tried to explain how our brain processes emotions. One of them is the classic subcortical route in which our limbic system plays a fundamental role. The type of melody influences recognition as happy or sad, and this recognition happens thanks to the inferior frontal gyrus, midline nuclear group and the anterior cingulate cortex.

Music capacity to produce such an intense pleasure and the stimulation it provides to the endogenous rewarding systems suggest that, if not essential, music it is still a great benefit for our mental and physical well-being.

A Cochrane review of 2015 evaluated the effects on listening to music for adults who suffered insomnia. 5 studies were included in the analysis (N = 264) to provide data about sleep quality on Pittsburgh Index, with results proving a benefit on listening to music. The effect was an increase in quality of sleep approximate to a standard deviation compared to no treatment or standard treatments. Only one study (N = 50, low quality evidence) showed data regarding latency at the beginning of the sleep cycle, total sleep time, sleep interruption and sleep efficacy. However it didn't show any evidence of improvement thanks to the music intervention. Authors concluded music can be effective to improve subjective quality of sleep in adults with insomnia. The intervention is safe and easy to administered, but more research is required to stablish the effects on other variables, as well as daytime consequences of insomnia.

A systematic review in 2018 regarding the possibility that music can improve quality of sleep in primary insomnia adults concluded that the improvement is only present with the relaxation that is associated to music, compared to the normal state of the patients.

This research is justified with the goal of evaluation in an objective way the quality of sleep in carers using the accelerometer, as well as subjective measures related to how listening to music can affect other sleeps variables (sleep interruptions, quality, total time, daytime consequences). The Cochrane review showed poor ratings of evidence in these variables except for quality of sleep being medium, as they were evaluated only in one study. High rating research is required to determine and establish the effect on daytime activity, which is why this clinical trial will take into account the authors recommendations to avoid bias. The use of the accelerometer will also provide data on physical activity in carers setting the ground for an intervention in the field.

Objectives

Main objective:

- To evaluate the effects of listening to music in sleep quality for oncology patients non-professional carers at home, and to evaluate the influence of specific factors that may modify that effect.

Secondary objectives:

* To assess the relationship between the waking state and the consequences during the day according to sleep characteristics. These include:

  3. Psychological results:

  1. Quality of life. 2. Carer overload. 4. Physical results:
  1. Sleepiness during the day.
  2. Physical activity, intensity and length evaluation.
* To assess carers satisfaction with the intervention.

Method:

Randomised clinical trail, single blinding carried out in several practices in the field of Primary Care of 6 units of Clinical Management belonging to the Malaga-Guadalhorce Health District, with informal carers of domiciliary oncological palliative patients.

Subject recruitment will be randomised and performed using a list of random numbers obtained using the program Epidat 3.1. This sample will take the oncological patients included in the Palliative Care Assistance Procedure showed on the Digital Clinical Records (DIRAYA) and having an informal care; every carer will be contacted and evaluated to the inclusion criteria, offering the possibility on taking part of the study if agreed and providing an informative leaflet. If accepted, a consent must be signed.

Randomising method will be as followed: several cards will be prepared labelled with "you have been included in the intervention group" or "you have been included in the control group", making equal numbers for the groups. They will be sealed on non-transparent envelopes, will be mixed and numbered after shuffling. The participants will be given a number (in order of acceptance to take part) and that number will be the assigned envelope and the group it contains. This procedure makes bias harder to occur.

Carers are offered the different groups and classified in intervention or control group, and this procedure it's performed by a sole person who will be responsible for randomising.

Once the researcher in charge of randomising knows the group the carer belongs to, he will proceed to inform them of the procedure the participants will be subject to without mentioning if they are intervention or control group so the patient will be oblivious.

This researcher will also inform the patient on how to use the accelerometer, the music program Spotify (Premium version) or the audio file through Google Drive (intervention or control group respectively).

Sample size: Based on data published by Jespersen et al. 201543 about quality of sleep the researchers are expecting to find an equivalent effect of medium standard differences of 0,776, with an alpha error of 0,05 and a beta error of 0,10. The sample size will be two groups of 35 patients (Epidat 3.1) increased to 40 to compensate for possible droppings/leaving.

Procedure for each group:

* Control group: The treatment will be performed according to what it is established in the Andalusian Palliative Care plan from the Health Council regarding carers, which include a complete initial evaluation regarding the 14 needs of Virginia Henderson, and the subsequent care plan and follow-up for problems or symptoms check; a basic health education for self-care and patient care will be administered, regarding feeding and hydration, physical exercise and leisure, medication, effective communication, skin care, prevention and treatment of constipation, and sleep hygiene. Carers from the control group will also receive the conventional health education that the carers will need to listen through headphones/earphones in the morning, using the mobile phone and the audio file shared in Google Drive, in daily sessions of 30 minutes during 7 days, while also wearing the accelerometer a week before and the week of the intervention. This way the caseload management nursing staff will be blinded on patient evaluation (see Masking and Randomising).
* Intervention group: carers will receive conventional health assistance complemented with music therapy with preselected music according to carers personal choice. The participants will have to listen to it half an hour before going to bed. The chosen music must be music that produces them pleasure or a nice feeling. This will be listened to via headphones/earphones and the mobile app Spotify (Premium version with free month trial). Daily session of 30 minutes during 7 days and the participants will wear the accelerometer the week before and the week of the intervention.

Statistical analysis:

A descriptive study will be performed with the collected variable using the medium and standard deviation in continuous normal variables, the confidence interval in punctual estimations; median and interquartile range in non-normal continuous variables, and frequency and percentages in categorical variables. The adjustment to normality will be determined with the Shapiro-Wilk test.

The basal values of both groups will be compared. Pre and post-intervention values will be analysed in both groups using the Student's t distribution for normal continuous variables and Wilcoxon's T for paired data in non-normal continuous variables. A multiple lineal regression will be also carried out where the dependant variable will be: self-perceived quality of sleep, total sleep time, total resting time, sleep interruption, sleep efficiency, quality of life, carer overload, daytime sleepiness, physical activity, intensity and length. The independent variables will be the intervention ones and the socio-demographic such as sex, age, education level, civil status, time dedicated to care, help received in care, time that the participants have been taking care of the patient, and relationship to person care for. The analysis will be similar for the use of painkillers, anxiolytic and sleeping pill medication.

The system developed for the PREDIMEDPLUS study will be used to process accelerometer data results. Processing and analysis of this data is also centralised, with an open source package, GGIR v. 1.5-1248 If statistically significant data are obtained in normal variables, the confidence intervals will be calculated at 95% to estimate values for the differences between the variables. The software to be used will be SPSS 23.0 and Epidat 3.01. Confidence interval will be 95% meaning only p values below 0,05 will be considered as statistically significant.

The present studio adjusts to the ethical recommendations:

1975 Helsinki Accords revised in 2013 (Ethical principles for research in humans (Helsinki, Adapted by the 64th General Assembly, Fortaleza, Brasil, October 2013).

All the personal information obtained in this study are confidential and will be dealt with in agreement to the EU 2016/679 regulation and the 27th of April 2016 GDPR (General Data Protection Regulation).

The 14th November 41/2002 law regulates the patient's autonomy and all the rights and duties regarding information and clinical records.

All the personal information collected in this study are confidential and will be treated in agreement with the 5th December 3/2018 Organic Law of Personal Data Protection and digital rights guarantee.

Participation is fully voluntary and an Informed consent will be signed to be admitted into the study.

ELIGIBILITY:
Inclusion Criteria:

* Being informal carer of a domiciliary palliative care patient.
* Having given informed consent to take part in the study.

Exclusion Criteria:

* Informal carer with severe hypoacusia, making it difficult to listen to the music on the phone/use of headphones
* Informal carer allergic to plastic and/or metal
* Informal carer with a programmed trip in the 2 weeks the study takes place
* Informal carer without mobile phone

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-02-12 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline quality of self-perceived sleep at 7 days through The Pittsburgh Sleep Quality Index (PSQI). | Pre-intervention/Post-intervention (0 and 7 days)
  Validated into Spanish. It values the sleep quality perceived by the subject. 7 different scores are obtained from the result, granting information for several components of the sleep quality: subjective quality, sleep latency, sleep duration, sleep efficiency, sleep disturbances (frequency of coughs, snores, heat, cold), sleeping pills intake, diurnal dysfunction (faculty to fall asleep through an activity because of tiredness). The sum of the scores in each component will be included into a Total Score (TS) from 0 to 21. According to Buysse and Cols, a TS of 5 will be the cutting point between a good and a bad sleep quality, less than 5 will show the presence of good sleep quality.
Change from baseline total sleep time and rest time (nighttime sleep and daytime rest / naps) at 7 days by accelerometry | Preintervention/Postintervention (0 and 7 days)
  The accelerometer triaxial: (GeneActiv, Activinsight Ltd, Kimbolton, Cambs, UK, http://www.geneactiv.org/). The data processing is done with an open source package in R, GGIR version 1.5-12.
Change from baseline sleep interruption level (number of awakenings and wakefulness after the onset of sleep) at 7 days by accelerometry | Preintervention/Postintervention ( 0 and 7 days)
  The accelerometer triaxial: (GeneActiv, Activinsight Ltd, Kimbolton, Cambs, UK, http://www.geneactiv.org/). The data processing is done with an open source package in R, GGIR version 1.5-12.
Change from baseline sleep efﬁciency (percentage of time in bed sleeping) (at the beginning and at 7 days) at 7 days by accelerometry. | Preintervention/Postintervention ( 0 and 7 days)
  The accelerometer triaxial: (GeneActiv, Activinsight Ltd, Kimbolton, Cambs, UK, http://www.geneactiv.org/). The data processing is done with an open source package in R, GGIR version 1.5-12.
Change from baseline levels of intensity of daily physical activity at 7 days by accelerometry. | Preintervention/Postintervention ( 0 and 7 days)
  The accelerometer triaxial: (GeneActiv, Activinsight Ltd, Kimbolton, Cambs, UK, http://www.geneactiv.org/). The data processing is done with an open source package in R, GGIR version 1.5-12.
Change from baseline daytime sleepiness at 7 days through the Epworth Sleepiness Scale (ESS). | Preintervention/Postintervention ( 0 and 7 days)
  Self-administered scale to measure diurnal sleepiness with 8 questions, scoring from 0 to 3 for a maximum score of 24. This scale is validated in Spanish.

SECONDARY OUTCOMES:
Change from baseline caregiver's effort index at 7 days through The Caregiver Strain Index Questionnaire (CSI) | Preintervention/Postintervention ( 0 and 7 days)
  Aimed to be answered by the caregiver of dependent people, containing 13 items with True/False answer. Every positive answer scores for 1. If the total is higher or equal to 7 it indicates a high level of strain. Being validated in Spanish, this is the scale used to evaluate the emotional and physical situation of the caregiver regarding their need to take care of a person in palliative care.
Change from baseline quality of life of the caregiver at 7 days through the EuroQol-5D-5L. | Preintervention/Postintervention ( 0 and 7 days)
  questionnaire validated in Spanish will be used, which describes health condition in 5 dimensions (mobility, personal care, day-to-day activities, pain/discomfort and anxiety/depression). It also present a visual analogue scale (VAS) graded 0 to 100 with the inserts "worst conceivable health condition" and "best conceivable health condition" in 0 and 100 respectively.
Client Satisfaction Questionnaire (CSQ-8) | Postintervention (7 days)
  8 questions answered through a Likert-type scale of 4 points and self-administered, with specific points to each item. The categories would be as follows: quality of the service, type of services, results and general satisfaction. It will include 3 open questions where the subjects answer what they liked most from the treatment, what they liked less, and what they would change. This tool has been proved to determine patient´s satisfaction with high reliability and coherence, being validated in the 8 items versions for Spanish speakers.
Socio-demographic carers data | Preintervention (0 days)
  : age, sex, civil status, education level, out-of-house job, time dedicated to care, help
  received for care, time that they have been taking care of someone, time the patient has
  been under palliative care, relationship with the patient, and consumption of painkillers, anxiolytic and sleeping pills medication.

CONTACTS AND LOCATIONS:
Overall Officials: Inmaculada Valero Cantero, Nurse, Principal Investigator — Distrito Sanitario Málaga- Guadalhorce. Servicio Andaluz de Salud; María Angeles Vázquez Sanchez, Doctor, Study Chair — University of Malaga; Yolanda Carrión Velasco, Nurse, Study Chair — Distrito Sanitario Málaga- Guadalhorce. Servicio Andaluz de Salud; Milagrosa Espinar Toledo, Nurse, Study Chair — Distrito Sanitario Málaga- Guadalhorce. Servicio Andaluz de Salud; Cristina Casals Sánchez, Doctor, Study Chair — University od Cádiz; Librado Valverde Velasco, Nurse, Study Chair — Distrito Sanitario Málaga- Guadalhorce. Servicio Andaluz de Salud; Milagros Reyes Sánchez, Nurse, Study Chair — Distrito Sanitario Málaga- Guadalhorce. Servicio Andaluz de Salud; Nuria Garcia-Agua Soler, Doctor, Study Chair — University of Malaga; Francisco Martínez Valero, chiropodist, Study Chair — National Health Service and Midlothian Foot Care, Dalkeith, Lothian, Scotland.; Francisco Javier Barón López, Doctor, Study Chair — University of Malaga; Jose Luís Casals Sánchez, Doctor, Study Chair — Hospital Universitario Virgen de la Victoria de Málaga; Ana Belén Arrabal Téllez, Nurse, Study Chair — Distrito Sanitario Axarquía-Este. Servicio Andaluz de Salud; Rosa Ana Serrano Benavente, doctor, Study Chair — Distrito Sanitario Axarquía-Este.Servicio Andaluz de Salud; Julia Wárnberg W, Doctor, Study Chair — University of Malaga
Locations (1):
- Inmaculada Valero Cantero, Málaga, Spain

REFERENCES:
- [Result] Cappuccio FP, Miller MA. Sleep and Cardio-Metabolic Disease. Curr Cardiol Rep. 2017 Sep 19;19(11):110. doi: 10.1007/s11886-017-0916-0. PMID 28929340
- [Result] Im E, Kim GS. Relationship between sleep duration and Framingham cardiovascular risk score and prevalence of cardiovascular disease in Koreans. Medicine (Baltimore). 2017 Sep;96(37):e7744. doi: 10.1097/MD.0000000000007744. PMID 28906359
- [Result] Komada Y, Nomura T, Kusumi M, Nakashima K, Okajima I, Sasai T, Inoue Y. A two-year follow-up study on the symptoms of sleep disturbances/insomnia and their effects on daytime functioning. Sleep Med. 2012 Oct;13(9):1115-21. doi: 10.1016/j.sleep.2012.05.015. Epub 2012 Jul 25. PMID 22841031
- [Result] Fu L, Jia L, Zhang W, Han P, Kang L, Ma Y, Yu H, Zhai T, Chen X, Guo Q. The association between sleep duration and physical performance in Chinese community-dwelling elderly. PLoS One. 2017 Mar 30;12(3):e0174832. doi: 10.1371/journal.pone.0174832. eCollection 2017. PMID 28358845
- [Result] Walsh JK. Clinical and socioeconomic correlates of insomnia. J Clin Psychiatry. 2004;65 Suppl 8:13-9. PMID 15153063
- [Result] Kotronoulas G, Wengstrom Y, Kearney N. Sleep patterns and sleep-impairing factors of persons providing informal care for people with cancer: a critical review of the literature. Cancer Nurs. 2013 Jan-Feb;36(1):E1-15. doi: 10.1097/NCC.0b013e3182456c38. PMID 22495497
- [Result] Harding R, Epiphaniou E, Hamilton D, Bridger S, Robinson V, George R, Beynon T, Higginson IJ. What are the perceived needs and challenges of informal caregivers in home cancer palliative care? Qualitative data to construct a feasible psycho-educational intervention. Support Care Cancer. 2012 Sep;20(9):1975-82. doi: 10.1007/s00520-011-1300-z. Epub 2011 Nov 10. PMID 22072049
- [Result] Dhruva A, Lee K, Paul SM, West C, Dunn L, Dodd M, Aouizerat BE, Cooper B, Swift P, Miaskowski C. Sleep-wake circadian activity rhythms and fatigue in family caregivers of oncology patients. Cancer Nurs. 2012 Jan-Feb;35(1):70-81. doi: 10.1097/NCC.0b013e3182194a25. PMID 21760489
- [Result] Lerdal A, Slatten K, Saghaug E, Grov EK, Normann AP, Lee KA, Bjorvatn B, Gay CL. Sleep among bereaved caregivers of patients admitted to hospice: a 1-year longitudinal pilot study. BMJ Open. 2016 Jan 4;6(1):e009345. doi: 10.1136/bmjopen-2015-009345. PMID 26729383
- [Result] Rittman M, Hinojosa MS, Findley K. Subjective sleep, burden, depression, and general health among caregivers of veterans poststroke. J Neurosci Nurs. 2009 Feb;41(1):39-52. doi: 10.1097/jnn.0b013e318193459a. PMID 19368070
- [Result] Gehrman P, Gooneratne NS, Brewster GS, Richards KC, Karlawish J. Impact of Alzheimer disease patients' sleep disturbances on their caregivers. Geriatr Nurs. 2018 Jan-Feb;39(1):60-65. doi: 10.1016/j.gerinurse.2017.06.003. Epub 2017 Jul 3. PMID 28684102
- [Result] Maltby KF, Sanderson CR, Lobb EA, Phillips JL. Sleep disturbances in caregivers of patients with advanced cancer: A systematic review. Palliat Support Care. 2017 Feb;15(1):125-140. doi: 10.1017/S1478951516001024. Epub 2017 Jan 18. PMID 28095943
- [Result] Reiner M, Niermann C, Jekauc D, Woll A. Long-term health benefits of physical activity--a systematic review of longitudinal studies. BMC Public Health. 2013 Sep 8;13:813. doi: 10.1186/1471-2458-13-813. PMID 24010994
- [Result] Lambert SD, Duncan LR, Kapellas S, Bruson AM, Myrand M, Santa Mina D, Culos-Reed N, Lambrou A. A Descriptive Systematic Review of Physical Activity Interventions for Caregivers: Effects on Caregivers' and Care Recipients' Psychosocial Outcomes, Physical Activity Levels, and Physical Health. Ann Behav Med. 2016 Dec;50(6):907-919. doi: 10.1007/s12160-016-9819-3. PMID 27439530
- [Result] Cuthbert CA, King-Shier K, Ruether D, Tapp DM, Culos-Reed SN. What is the State of the Science on Physical Activity Interventions for Family Caregivers? A Systematic Review and RE-AIM Evaluation. J Phys Act Health. 2017 Jul;14(7):578-595. doi: 10.1123/jpah.2016-0280. Epub 2017 Mar 14. PMID 28290737
- [Result] Hirano A, Suzuki Y, Kuzuya M, Onishi J, Ban N, Umegaki H. Influence of regular exercise on subjective sense of burden and physical symptoms in community-dwelling caregivers of dementia patients: a randomized controlled trial. Arch Gerontol Geriatr. 2011 Sep-Oct;53(2):e158-63. doi: 10.1016/j.archger.2010.08.004. Epub 2010 Sep 17. PMID 20850878
- [Result] King AC, Baumann K, O'Sullivan P, Wilcox S, Castro C. Effects of moderate-intensity exercise on physiological, behavioral, and emotional responses to family caregiving: a randomized controlled trial. J Gerontol A Biol Sci Med Sci. 2002 Jan;57(1):M26-36. doi: 10.1093/gerona/57.1.m26. PMID 11773209
- [Result] DeMartinis NA, Kamath J, Winokur A. New approaches for the treatment of sleep disorders. Adv Pharmacol. 2009;57:187-235. doi: 10.1016/S1054-3589(08)57005-0. Epub 2009 Nov 27. PMID 20230762
- [Result] Schroeck JL, Ford J, Conway EL, Kurtzhalts KE, Gee ME, Vollmer KA, Mergenhagen KA. Review of Safety and Efficacy of Sleep Medicines in Older Adults. Clin Ther. 2016 Nov;38(11):2340-2372. doi: 10.1016/j.clinthera.2016.09.010. Epub 2016 Oct 15. PMID 27751669
- [Result] Wilt TJ, MacDonald R, Brasure M, Olson CM, Carlyle M, Fuchs E, Khawaja IS, Diem S, Koffel E, Ouellette J, Butler M, Kane RL. Pharmacologic Treatment of Insomnia Disorder: An Evidence Report for a Clinical Practice Guideline by the American College of Physicians. Ann Intern Med. 2016 Jul 19;165(2):103-12. doi: 10.7326/M15-1781. Epub 2016 May 3. PMID 27136278
- [Result] Mercier J, Savard J, Bernard P. Exercise interventions to improve sleep in cancer patients: A systematic review and meta-analysis. Sleep Med Rev. 2017 Dec;36:43-56. doi: 10.1016/j.smrv.2016.11.001. Epub 2016 Nov 10. PMID 27939642
- [Result] van Straten A, van der Zweerde T, Kleiboer A, Cuijpers P, Morin CM, Lancee J. Cognitive and behavioral therapies in the treatment of insomnia: A meta-analysis. Sleep Med Rev. 2018 Apr;38:3-16. doi: 10.1016/j.smrv.2017.02.001. Epub 2017 Feb 9. PMID 28392168
- [Result] Davidson RJ, Irwin W. The functional neuroanatomy of emotion and affective style. Trends Cogn Sci. 1999 Jan;3(1):11-21. doi: 10.1016/s1364-6613(98)01265-0. PMID 10234222
- [Result] Peretz I, Gagnon L, Bouchard B. Music and emotion: perceptual determinants, immediacy, and isolation after brain damage. Cognition. 1998 Aug;68(2):111-41. doi: 10.1016/s0010-0277(98)00043-2. PMID 9818509
- [Result] Mizuno T, Sugishita M. Neural correlates underlying perception of tonality-related emotional contents. Neuroreport. 2007 Oct 29;18(16):1651-5. doi: 10.1097/WNR.0b013e3282f0b787. PMID 17921862
- [Result] Soria-Urios G, Duque P, Garcia-Moreno JM. [Music and brain: neuroscientific foundations and musical disorders]. Rev Neurol. 2011 Jan 1;52(1):45-55. Spanish. PMID 21246493
- [Result] Blood AJ, Zatorre RJ. Intensely pleasurable responses to music correlate with activity in brain regions implicated in reward and emotion. Proc Natl Acad Sci U S A. 2001 Sep 25;98(20):11818-23. doi: 10.1073/pnas.191355898. PMID 11573015
- [Result] Jespersen KV, Koenig J, Jennum P, Vuust P. Music for insomnia in adults. Cochrane Database Syst Rev. 2015 Aug 13;2015(8):CD010459. doi: 10.1002/14651858.CD010459.pub2. PMID 26270746
- [Result] Feng F, Zhang Y, Hou J, Cai J, Jiang Q, Li X, Zhao Q, Li BA. Can music improve sleep quality in adults with primary insomnia? A systematic review and network meta-analysis. Int J Nurs Stud. 2018 Jan;77:189-196. doi: 10.1016/j.ijnurstu.2017.10.011. Epub 2017 Oct 23. PMID 29100201
- [Derived] Valero-Cantero I, Carrion-Velasco Y, Casals C, Martinez-Valero FJ, Baron-Lopez FJ, Vazquez-Sanchez MA. Intervention to improve quality of sleep of palliative patient carers in the community: protocol for a multicentre randomised controlled trial. BMC Nurs. 2020 Nov 16;19(1):107. doi: 10.1186/s12912-020-00501-2. PMID 33292183
- See also: World Health Organization. Global Recommendations on Physical Activity for Health. [Libro en Internet] Génova (Suiza). OMS; 2010. [acceso 25 de marzo de 2018]. — http://www.who.int/dietphysicalactivity/publications/9789241599979/en/
- See also: Andalusian Palliative Care Plan — https://www.juntadeandalucia.es/organismos/saludyfamilias/areas/planificacion/planes-integrales/paginas/pacpa.html